CLINICAL TRIAL: NCT06751199
Title: Investigation of Dose Escalation and Dose Expansion Study on the Safety and Efficacy of Allogeneic Human Umbilical Cord Mesenchymal Stem Cells Combined With Allogeneic Islet Transplantation for the Treatment of Diabetes
Brief Title: UCMSCs Combined With Allogeneic Islet Transplantation for the Treatment of Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZYZ-CTIM-2023-IIT
Record Dates: First submitted 2024-10-10; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): allogeneic islet combined with hUCMSCs
  Interventions: Drug: human umbilical cord mesenchymal stem cells; Drug: allogeneic islet
- Comparator (Active Comparator): allogeneic islet
  Interventions: Drug: allogeneic islet

INTERVENTIONS:
Drug: human umbilical cord mesenchymal stem cells — Portal vein infusion human umbilical cord mesenchymal stem cells
  Arms: Experimental
Drug: allogeneic islet — Portal vein infusion of allogeneic islet

SUMMARY:
The aim is to Investigate the safety and efficacy of Portal vein infusion Allogeneic Human umbilical cord mesenchymal stem cells combined with Allogeneic islet transplantation for the treatment of diabetes

DETAILED DESCRIPTION:
This is an investigator-initiated trial (IIT). The first part is an open-label, dose-escalation study involving 9 patients between the ages of 18 and 70. The second part is a non-randomized, active comparator-controlled IIT with a parallel design, comparing allogeneic islet transplantation combined with human umbilical cord mesenchymal stem cells (hUCMSCs) to allogeneic islet transplantation alone in patients with diabetes.Besides safety, preservation of endogenous insulin production (measured as C-peptide concentrations) together with metabolic control, diabetes treatment satisfaction and immunological profile will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the 1999 World Health Organization diagnostic criteria for diabetes.
2. Aged 18-70, no gender restriction.
3. Islet function failure: fasting C-peptide < 0.1 nmol/L, 2-hour postprandial C-peptide < 0.2 nmol/L, and HbA1c ≥ 7%.
4. Meets the indications for islet transplantation alone:

   i. Type 1 diabetes patients who experience unstable blood glucose despite strict insulin therapy, including frequent hypoglycemia or at least one severe hypoglycemic event in the past 12 months, or those with serious complications in other organs such as the kidneys; ii. Type 2 diabetes progressing to islet failure with poor blood glucose control as described above; iii. Patients with chronic pancreatitis or non-malignant pancreatic tumors who have undergone total or near-total pancreatectomy may receive autologous islet transplantation concurrently or allogeneic islet transplantation later.
5. The patient and their family or legal guardian voluntarily consent to stem cell transplantation therapy and sign the informed consent form.

Exclusion Criteria:

1. Diabetic ketoacidosis that is not yet controlled.
2. Severe allergic constitution, meaning prone to allergic reactions without a clear and identifiable cause.
3. BMI < 14 or > 35.
4. Severe anemia (hemoglobin < 8 g/dL in males, < 7 g/dL in females).
5. HIV-positive, carriers of viral hepatitis or in the active phase, or other uncontrolled infectious diseases.
6. History of acute pancreatitis, pulmonary embolism, or other thrombotic diseases, as well as severe heart, liver, kidney, respiratory, or neurological diseases.
7. Patients with gestational diabetes, monogenic diabetes, diabetes due to pancreatic damage, or other secondary diabetes (e.g., diabetes caused by Cushing's syndrome, thyroid dysfunction, or acromegaly).
8. Pregnant women or those planning pregnancy within 3 months before or after treatment, and women who are breastfeeding.
9. Patients with mental illness, alcohol or drug abuse, who are unable to cooperate with treatment.
10. Known or suspected tumors.
11. History of other autoimmune diseases or hematological disorders.
12. Any other clinical conditions that, in the investigator's judgment, may pose a risk to the participant's safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety assessment: Registration of adverse events | Throughout the study until Week 52
  Changes in safety parameters of patients during the study period since baseline. Measured through the registration of adverse events.
Efficacy Assessment: Evaluation of islet function | Throughout the study until Week 52
  Change of C-peptide Area Under the Curve (AUC) (0-120 min) for Mixed Meal Tolerance Test (MMTT) at Week 52 compared to test performed before start of treatment.

SECONDARY OUTCOMES:
Efficacy Assessment: HbA1c | Week 52
  Changes in patient HbA1c levels from baseline during the study period
Dose of exogenous insulin | Week 52
  Changes in daily exogenous insulin requirements during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yin, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided